CLINICAL TRIAL: NCT04154683
Title: Diagnostic Performance of Optical Biopsy by Cellvizio® in Gynecological Surgery
Brief Title: Optical Biopsy in Gynecological Surgery
Acronym: GYNECOPTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0945; 2019-A01724-53 (Other: ID-RCB)
Record Dates: First submitted 2019-11-05; First posted 2019-11-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Surgical Procedures
Keywords: salpingectomy; Cellvizio®; optical biopsy; unilateral or bilateral salpingectomy; ovariectomy; Endometriosis; surgery for cervical; ovarian cancer
MeSH Terms: conditions — Endometriosis; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group using Cellvizio® optical biopsy (Experimental)
  Interventions: Device: Cellvizio®

INTERVENTIONS:
Device: Cellvizio® — use of the Cellvizio® optical biopsy

SUMMARY:
Optical biopsy is a new technology that generates a real-time, cell-based, high-resolution view and analysis of tissues. Observation is instantaneous and non-invasive. This allows reliable and fast diagnosis which facilitates decision making as well as patient management.

The investigator have already conducted a feasibility study on the use of this new technology to evaluate ovarian and tubal pre-cancerous lesions in laparoscopy. In this new study, he wants to continue investigations, expand its use to other gynecological pathologies, and demonstrate the benefit of such a non-invasive technology in gynecology on the one hand in the diagnosis of lesions but also to appreciate the margins as accurately as possible surgical excision of tumors and / or endometriosis lesions.

The investigator have set up a prospective monocentric descriptive study. The hypothesis is that optical biopsy by Cellvizio® allows to observe in real time microscopically tissues and to characterize them in the field of gynecological surgery

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or more
* Informed and signed consent
* Planned surgery under laparoscopy and included in the list below:

  * unilateral or bilateral salpingectomy
  * hysterectomy
  * ovariectomy
  * surgery of endometriosis
  * surgery for cancer of the cervix, endometrium, ovaries

Exclusion Criteria:

* Interview revealing disorder entailing unacceptable risk of postoperative complications: coagulation disorder, immune system disorder, evolutive disease, etc.
* Pregnancy or desire of pregnancy during the study period, breastfeeding
* Hypersensitivity to Fluorescein or any of its excipients
* History of life-threatening reaction during angiography
* Known allergic reactions and hypersensitivity
* Severe asthma, heart and / or lung disease, diabetes
* Person on beta-blocker treatment
* Inability to understand information provided
* Not covered by a national health insurance scheme, prisoner or under administrative supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
correlation optical biopsy and anatomopathology | day 0
  The interpretation of the results of the optical biopsy will be compared with the interpretation of the pathological results for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Gautier CHENE, MD, Principal Investigator — Gynaecology Department, Hôpital Femme Mère Enfant Hospices Civils de Lyon
Locations (2):
- France (2):
  - Gynaecology Department, Hôpital Femme Mère Enfant Hospices Civisl de Lyon, Bron
  - Service de Gynécologie, HFME, Hospices Civils de Lyon, Bron